CLINICAL TRIAL: NCT07404150
Title: Women, Weight, and Well-Being: An Observational Study of an Interdisciplinary Lifestyle Program With or Without GLP-1 Therapy to Support Intentional Weight Loss, Reduce Internalized Weight Bias, and Improve Positive Health Behaviors in Women With Obesity-Related Cardiovascular Risk
Brief Title: Women, Weight, and Well-being
Status: Enrolling by invitation | Type: Observational
Sponsor: Heather Conradson (Other)
Collaborators: Symphony of Health Connections (Other); Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Heather Conradson, Principal Investigator, Nurse Scientist (PhD, RN), Symphony of Health Connections
Organization: Symphony of Health Connections (Other)
Other Study IDs: HREBA-Protocol-CHC 25-00092
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity and Cardiovascular Risk
Keywords: obesity; women; cardiovascular risk
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women aged 35-75 years whose weight poses a CVD risk: Eligibility includes BMI ≥ 30 kg/m² with waist circumference > 88 cm, or BMI ≥ 27 kg/m² with obesity-related health conditions consistent with Edmonton Obesity Staging System (EOSS) stage 1 or higher. Participants take part in a 12-month, women-focused lifestyle program delivered in groups, with added individual support. The program includes 21 group classes over 12 months, plus brief check-ins every two weeks for the first 6 months and then monthly until 12 months. Sessions focus on practical, sustainable changes related to nourishment (not restrictive dieting), intentional movement for health, and emotional well-being (e.g., self-compassion skills, sleep support, and mindfulness or meditation strategies). The program emphasizes the biology of weight gain and provides support in a stigma-free, non-judgmental way. Some participants may also use GLP-1 medication as part of their usual medical care.
  Interventions: Other: lifestyle change program

INTERVENTIONS:
Other: lifestyle change program — 21 Group classes provided by interdisciplinary team (RN,RD,KIN); BI-weekly individual follow-up for first 6 months then monthly in addition to classes

SUMMARY:
Women, Weight and Well-Being is a 12-month research study looking at how a supportive lifestyle program may help women whose weight increases their risk for heart disease.

We want to understand whether taking part in the program is linked with changes in: body weight and waist size; blood pressure and bloodwork related to heart health (such as cholesterol and A1C); health habits (movement, eating patterns, sleep); well-being and how women feel about their bodies, including the effects of weight stigma.

About 60 women aged 35-75 will take part. Participants will attend group sessions and have one-on-one support from a nurse, dietitian, and kinesiologist. Some participants may also use GLP-1 medication (a type of medication that can support weight loss) as part of their regular medical care, if it is right for them. The study does not assign medication. We simply observe outcomes over time.

Information will be collected at the start of the program, at 6 months, and at 12 months using measurements (such as weight, waist, blood pressure), routine lab results, and questionnaires about health and well-being.

DETAILED DESCRIPTION:
Women with obesity face a higher risk of cardiovascular disease and cardiometabolic complications, yet this risk is frequently under addressed, creating a gap in cardiovascular care. Compounding this risk are the psychological impacts of weight stigma, internalized weight bias (IWB), the internal adoption of society's negative stereotypes about body weight, which is more prevalent among women and linked to chronic stress, healthcare avoidance, disruptions in health-promoting behaviours, and increased morbidity and mortality.

A 12-month observational study has been designed to address these gaps by offering and assessing the impact of an interdisciplinary lifestyle program on weight loss, cardiovascular, and psychological outcomes in women whose weight poses a cardiovascular disease (CVD) risk. It integrates medical, nutritional, exercise and psychological support through group-based education, individualized care, and the option to use GLP-1 therapy. The program offers stigma-free, relationship-centred support grounded in the biology of adiposity and the importance of self-compassion, nourishing and non-restrictive nutrition, movement, sleep, and emotional well-being.

This study will enroll 60 women aged 35-75 years whose weight poses a CVD risk. Eligibility includes BMI ≥ 30 kg/m² with waist circumference >88 cm or BMI ≥ 27 kg/m² obesity-related health conditions consistent with Edmonton Obesity Staging System Stage ≥ 1. Participants may choose a lifestyle-only approach or add GLP-1 therapy, with nurse-led titration and monitoring.

The program includes three phases: Phase 1 (Weeks 0 to 6) offers weekly group sessions and individual visits; Phase 2 (Weeks 7 to 24) provides biweekly sessions and a midpoint assessment; and Phase 3 (Months 7 to 12) delivers monthly support and long-term follow-up. Collaborating with the participant's cardiologist or primary care provider, an interdisciplinary team (RN, RD, Kinesiologist) will provide group and one-on-one support. RN or RD check-ins occur biweekly during the first six months and monthly thereafter, with RN-led support for medication titration as needed.

Data including weight, waist circumference, BP, lipids, HbA1C, exercise capacity (DASI, grip strength, BODY-Q physical function), dietary patterns (24hr Dietary Recall, Mediterranean Diet Score, BODY-Q dietary behavior), food noise (FNQ), psychological well-being (PERMA, EQ-5D-5L, BODY-Q social function, Psychological function, SCS-SF), sleep (STOP-BANG) and internalized weight bias (WBIS) will be collected at baseline, 6, and 12 months. Focus groups will explore participant experience. The findings will inform women-centred care by evaluating whether this interdisciplinary program promotes positive health behaviours, enhances well-being, and improves cardiometabolic risk.

ELIGIBILITY:
Inclusion Criteria:

* • Ability to provide informed consent before any study-related activities

  * Female
  * Age between 35 and 75 years
  * BMI ≥ 30 kg/m² with waist circumference ≥ 88 cm or BMI ≥ 27 kg/m² with obesity-related health conditions consistent with Edmonton Obesity Staging System Stage ≥ 1.
  * Willingness to engage in a 12-month interdisciplinary lifestyle program
  * Ability to attend group sessions (in person or virtually) and complete follow-up visits
  * Alberta resident with Alberta Health Care insurance
  * Sufficient proficiency in English to engage with group material and communications

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during the study period

  * Diagnosis of type 1 diabetes
  * Life-limiting illness or severe medical condition where weight loss would not be clinically appropriate (e.g., advanced cancer, end-stage organ failure); clinical judgment will be used to assess suitability
  * Severe psychiatric illness or cognitive impairment that would interfere with participation in group sessions or study procedures
  * Current participation in another weight management or investigational study
  * Inability to comply with study procedures due to logistical, medical, or language barriers

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 35-75 years whose weight poses a CVD risk.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-06-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Percent weight change and internalized weight bias (WBIS) | 18 months
  In addition to weight change we will measure , waist circumference, BP, lipids, HbA1C, exercise capacity (DASI, grip strength, BODY-Q physical function), dietary patterns (24hr Dietary Recall, Mediterranean Diet Score, BODY-Q dietary behavior), food noise, psychological well-being (PERMA, EQ-5D-5L, BODY-Q social function, Psychological function, SCS-SF), sleep (STOP-BANG) will be collected at baseline, 6, and 12 months. Focus groups will explore participant experience.

CONTACTS AND LOCATIONS:
Locations (1):
- Symphony of Health Connections, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No